CLINICAL TRIAL: NCT00867061
Title: A Phase 1/2, Single-Arm Study To Assess The Efficacy and Safety Of 5-day Continuous Intravenous Dosing Of ON 01910.Na Administered Every 2 Weeks in Patients With Intermediate-1, Intermediate-2, or High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Efficacy and Safety of 5-day Dosing of ON 01910.Na in Intermediate-1,-2, or High Risk Myelodysplastic Syndrome (MDS)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Mutual decision by site and sponsor because of difficulty recruiting Patients.
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-11
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic; IPSS Intermediate 1; IPSS Intermediate 2; IPSS High risk
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ON 01910.Na Concentrate — 5-day continuous intravenous dosing of ON 01910.Na given every 2 weeks (1 cycle) at a dose of 800 mg/m2/day or 1500mg/m2/day for up to 24 cycles.

SUMMARY:
For MDS patients who have not responded to or have progressed after an initial response to DNA methyltransferase inhibitors (DNMTI) and are not stem cell transplant candidates, therapeutic options are limited. Participation in clinical trials such as this one may be considered. The specific objectives of this trial are to find out which dose of ON 01910.Na can be safety given to MDS patients and then find out if this dose of drug has any beneficial effects on the patients' disease. ON 01910.Na is a new, experimental drug; the reason for doing this trial is based on the anti-cancer activity of ON 01910.Na that has been observed in laboratory experiments and in early clinical trials.

DETAILED DESCRIPTION:
This is a single center, open label, phase 1/2 study in which two to thirty three patients with Intermediate-1, Intermediate-2, or High risk MDS will receive ON 01910.Na as a intravenous continuous infusion (IVCI) over 24 hours for 5 consecutive days every 2 weeks.

In the phase 1 component of this trial the maximum tolerated dose of ON1910.Na in patients with Intermediate-1, Intermediate-2 or High Risk myelodysplastic syndromes will be determined. A standard "3+3" dose escalation scheme will be followed with up to six patients treated at the 800 mg/m2/day dose level. Patients will be observed for 2 cycles before dose escalation occurs. If none of the initial three patients in the 800 mg/m2/day cohort experience dose-limiting toxicity (DLT), during the first two cycles, then a new cohort of three patients will be treated at the 1500 mg/m2/day dose level. If none of the initial three patients in the 1500 mg/m2/day cohort experience DLT during the first two cycles, three additional patients will be treated at the 1500 mg/m2/day level. If no more than one of the six patients at the 1500 mg/m2/day dose level experiences a DLT, then that dose level will be confirmed as the MTD and no further dose escalation will occur.

If one of the three patients in the 800 mg/m2/day cohort experiences DLT during the first two cycles, then up to three additional patients will be treated at the same dose level. Escalation to 1500 mg/m2/day will proceed if only one of the six patients experiences DLT at the 800 mg/m2/day dose level. If two or more patients in the 800 mg/m2/day cohort experience DLT during the first two cycles, then the maximum tolerated dose (MTD) will have been exceeded, no further dose escalation will occur, and a full safety review will determine if further enrollment of patients will proceed.

If the 800 mg/m2/day dose level is under consideration as the MTD (i.e. if ≥ 2 patients experience DLT at the 1500 mg/m2/day dose level), and only three patients were treated before escalation to 1500 mg/m2/day, then three additional patients will be accrued. If no more than one of the six patients at the 800 mg/m2/day dose level experiences a DLT, then that dose level will be confirmed as the MTD.

Once the phase 1 portion of the study is completed, accrual to the phase 2 portion will begin. Patients treated at the MTD during the phase 1 portion will be included in the phase 2 component and will be evaluated for response and secondary end points.

The total study duration is 29 weeks, which includes a 2-week screening phase, a 23-week dosing phase, and a 4-week follow-up phase that begins after the last dose of ON 01910.Na. Patients will be assessed for response and will undergo follow up.

Patients who drop out for any reason will not be replaced. Patients who achieve a complete or partial response or stabilization of their disease by week 25 are eligible to receive an additional 24 weeks of ON 01910.Na at the same dose they received during the first 24 weeks of treatment(800 or 1500 mg/m2/day IVCI for 5 days Q2W).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS confirmed within 4 weeks prior to study entry according to the World Health Organization (WHO) Criteria or the French-American-British (FAB) Classification.
* IPSS score of at least 0.5 (Intermediate-1, Intermediate-2 or High Risk MDS)
* Failure of, or insufficient response to 5-azacitidine or decitabine administered for 4 to 6 cycles.
* Failed to respond to, relapsed following, or opted not to participate in bone marrow transplantation.
* Off all other treatments for MDS, including filgrastim (G-CSF) and erythropoietin for at least 2 weeks, and off standard or investigational MDS therapies for four weeks.
* ECOG Performance Status 0, 1 or 2.
* Adequate contraceptive [including prescription oral contraceptives (birth control pills), contraceptive injections, intrauterine device (IUD), double-barrier method (spermicidal jelly or foam with condoms or diaphragm), contraceptive patch, or surgical sterilization] before entry and throughout the study for female patients of reproductive potential.
* Female patients with reproductive potential must have a negative serum beta-HCG pregnancy test at screening.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Patient (or his/her legally authorized representative) must have signed an informed consent document indicating that he/she understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

* Anemia due to factors other than MDS (including hemolysis or gastrointestinal bleeding).
* Hypoplastic MDS (cellularity <10%).
* Any active malignancy within the past year except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast.
* History of HIV-1 seropositivity.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Active infection not adequately responding to appropriate therapy.
* Total bilirubin ≥ 1.5 mg/dL not related to hemolysis or Gilbert's disease, ALT or AST ≥ 2 X ULN.
* Serum creatinine ≥ 1.5 mg/dL or calculated creatinine clearance ≤ 60 ml/min/1.73 m2
* Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <134 Meq/L).
* Female patients who are pregnant or lactating.
* Male patients with female sexual partners who are unwilling to follow the strict contraception requirements described in this protocol.
* Major surgery without full recovery or major surgery within 3 weeks of ON 01910.Na treatment start.
* Uncontrolled hypertension (defined as a systolic pressure ≥ 160 and/or a diastolic pressure ≥ 110).
* New onset seizures (within 3 months prior to the first dose of ON 01910.Na) or poorly controlled seizures.
* Any concurrent investigational agent or chemotherapy, radiotherapy or immunotherapy.
* Treatment with myeloid growth factors or erythropoiesis stimulating agents (ESA) within 2 weeks of starting ON 01910.Na.
* Treatment with standard MDS therapies or investigational therapy within 4 weeks of starting ON 01910.Na.
* Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (in Phase 1) | 1 month
Response according to International Working Group criteria (in Phase 2) | 2 to 3 months

SECONDARY OUTCOMES:
Response time | 2 - 6 months
IPSS score | 2 to 6 months
Neutrophil response | 2 to 6 months
Platelet response | 2 to 6 months
Erythroid response | 2 to 6 months
Overall survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Klimek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Background] Jimeno A, Chan A, Cusatis G, Zhang X, Wheelhouse J, Solomon A, Chan F, Zhao M, Cosenza SC, Ramana Reddy MV, Rudek MA, Kulesza P, Donehower RC, Reddy EP, Hidalgo M. Evaluation of the novel mitotic modulator ON 01910.Na in pancreatic cancer and preclinical development of an ex vivo predictive assay. Oncogene. 2009 Jan 29;28(4):610-8. doi: 10.1038/onc.2008.424. Epub 2008 Nov 24. PMID 19029951
- [Background] Cheson BD, Bennett JM, Kantarjian H, Pinto A, Schiffer CA, Nimer SD, Lowenberg B, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Wijermans PW, Gore S, Greenberg PL; World Health Organization(WHO) international working group. Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood. 2000 Dec 1;96(12):3671-4. PMID 11090046
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Aarthi Shenoy, Loretta Pfannes, Francois Wilhelm, Manoj Maniar, Neal Young, and Elaine M Sloand Suppression of Cyclin D 1 (CD1) by ON 01910.Na Is Associated with Decreased Survival or Trisomy 8 Myelodysplastic Bone Marrow: A Potential Targetted Therapy for Trisomy 8 MDS. Blood (ASH Annual Meeting Abstracts), Nov 2008; 112: 1651.
- [Background] Elaine M. Sloand, Loretta Pfannes, Ramana Reddy, Premkumar Reddy, Jerome S. Groopman, and Neal S. Young Suppression of Cyclin D1 by ON 01910.Na Is Associated with Decreased Survival of Trisomy 8 Myelodyplastic Bone Marrow Progenitors: A Potential Targetted Therapy. Blood (ASH Annual Meeting Abstracts), Nov 2007; 110: 822.
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- See also: Website of trial study center. Provides cancer care information to healthcare professionals, researchers, patients, family members, and the public. — http://www.mskcc.org